CLINICAL TRIAL: NCT00774878
Title: Multicenter, Randomized, Open Label Study Evaluating an Anti Insulin-like Growth Factor-1 Receptor (IGF-1R/CD221) Monoclonal Antibody, AVE1642, Administered Every 4 Weeks in Combination With Fulvestrant (Faslodex®) in Postmenopausal Patients With Advanced Hormono-dependent Breast Cancer
Brief Title: Study of AVE1642 (IGF-1R/CD221) in Combination With Fulvestrant (Faslodex®) in Postmenopausal Patients With Advanced Hormono-dependent Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue the AVE1642 development program, not due to any safety or efficacy concerns
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD10631; EudraCT Number: 2008-000810-54
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Breast Tumors; Anti IGF-1R; Hormonosensitivity
MeSH Terms: conditions — Breast Neoplasms | interventions — AVE1642; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: AVE1642; Drug: Fulvestrant
- Arm B (Active Comparator)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: AVE1642 — AVE1642 is administered intravenously at the dose of 8 mg/kg.
  Arms: Arm A
Drug: Fulvestrant — Fulvestrant is administered as a slow intramuscular injection (just before the AVE1642 infusion when given in combination).

SUMMARY:
The purpose of this study is to evaluate the clinical activity of AVE1642 in combination with fulvestrant and of fulvestrant alone in terms of clinical benefit as the rate of "complete response", "partial response" and "stabilization of the disease".

The additional objectives are to evaluate the safety profile of AVE1642 in combination with fulvestrant and of fulvestrant alone, to assess the rate of patients without disease progression at 6 months and the overall progression-free survival time. An evaluation of the pharmacokinetics and pharmacodynamics interactions between AVE1642 and fulvestrant will also be performed.

The biological activity of treatment will be assessed on tumor biopsies, when possible The potential immunogenicity of AVE1642 will be studied

DETAILED DESCRIPTION:
The study treatment will be administered until disease progression, unacceptable toxicity or patient willingness to discontinue.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* Aromatase inhibitor as the last hormonal treatment
* Breast adenocarcinoma with positive hormone receptor
* Measurable disease as per RECIST definition

Exclusion Criteria:

* ECOG performance status (PS) > 2
* Prior exposure to fulvestrant or to an anti IGF-1R compound
* No evidence of hormonosensitivity
* HER 2-neu positive tumor
* More than one prior regimen of chemotherapy for metastatic disease

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Clinical benefit defined as a confirmed complete response (CR) or a confirmed partial response (PR) or a stable disease (SD)lasting at least 24 weeks (6 cycles) | 6 cycles

SECONDARY OUTCOMES:
Progression Free rate | at 6 months
Safety (TEAEs, hematology, biochemistry parameters) | study period

CONTACTS AND LOCATIONS:
Overall Officials: Henri ROCHE, Professor, Principal Investigator — Institut Claudius Regaud (TOULOUSE - FRANCE)
Locations (3):
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Barcelona, Spain